CLINICAL TRIAL: NCT04176692
Title: The Movement Pattern of Shoulder Complex and the Intervention Effects of Therapeutic Exercise in Patients With Proximal Humerus Fracture
Brief Title: The Effects of Muscle Characteristics on the Control of Shoulder Complex During Functional Movements
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Po-Tsun Chen, Principal Investigator, Tzu Chi University
Other Study IDs: MOST108-2314-B-320 -001-
Record Dates: First submitted 2019-11-16; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Other Instability of Joint, Shoulder Region; Strain of Shoulder Muscle (Disorder); Movement Disorders
Keywords: scapula dyskinesia; muscle stiffness; scapulohumeral rhythm; electromyography
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The movement control of shoulder joint relies not only on the glenohumeral joint, but also the critical contributions from scapulothoracic joint. The relating scapula muscle strength, scapula mobility and, the most important of all, the capacity of neuromuscular control should be integrated into the rehabilitation program for patients with shoulder disorders. With regarding to the subacromial impingement syndrome or rotator tendinopathy, the status of scapula dyskinesia and dysfunctions were improved significantly after the intervention of scapula-emphasized exercise. But there was no study addressed the relationships between stiffness of relating muscles and the deficits of scapula movement. The stiffness had been shown to serve an important role in functional performance of the corresponding joint. For example, the decreased elasticity of supraspinatus muscle was noticed on affected side comparing in patients with impingement syndrome.Few studies examined the effects of altered muscle stiffness on kinematic performance in shoulder complex. Laudner et al. found that the stiffer the latismuss dorsi muscle was, the less upward rotation and posterior tilting, and the more internal rotation of scapula during arm elevation was exhibited in asymptomatic swimmers. Another study showed that the increased range of external rotation and posterior tilt of scapula during arm elevation were associated with the decreased stiffness of pectoralis minor. The recent study presented that the electromyographic activities and elasticities of middle deltoid, supraspinatus, and infraspinatus muscles correlated significantly with the tissue elasticity during shoulder movement in healthy shoulder. However, there was no scientific information directly to prove the changes in characteristics of rotator cuff function as well as the impacts on kinematic control of shoulder complex. Therefore, the aim of this study is to examine the relationship among characteristics of muscle properties and kinematic control healthy swimmers.

ELIGIBILITY:
Inclusion Criteria:

* freestyle swimmers with health shoulders

Exclusion Criteria:

* the past or current shoulder pain or disorders are examined by history taking and screening tests: shoulder impingement syndrome, instability, bony deformity, trauma, nerve injury or entrapment.

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: adolescent swimmers in junior or senior high school swimming team with regular training
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
scapulohumeral kinematics | through study completion, an average 11 months
  the three-dimensional movements of humerus-to-trunk and scapula-to-trunk motions (degree) measured by the electromagnetic motion capture system
muscle activities | through study completion, an average 11 months
  muscle activitiy of upper trapezius, middle deltoid, serratus anterior, infraspinatus, lower trapezius recorded by the surface electromyography

SECONDARY OUTCOMES:
muscle strength | through study completion, an average 11 months
  maximum muscle strength of upper trapezius, middle deltoid, serratus anterior, lower trapezius, internal and external rotators recorded by the hand-held dynamometer
muscle stiffness | through study completion, an average 11 months
  muscle stiffness of upper trapezius, middle deltoid, serratus anterior, infraspinatus, lower trapezius recorded by the tissue-hardness measurement device

CONTACTS AND LOCATIONS:
Overall Officials: Po-Tsun Chen, Principal Investigator — Tzu Chi University
Locations (1):
- Tzu Chi University, Hualien City, 請選擇, Taiwan

IPD SHARING:
Plan to Share IPD: No